CLINICAL TRIAL: NCT03427242
Title: A Phase II Study of Apatinib Treatment for Advanced Biliary Tract Carcinoma After Failure of the First-line Chemotherapy
Brief Title: Apatinib for Advanced Biliary Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, MD, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDZL-BTA
Record Dates: First submitted 2018-01-25; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2017-11

CONDITIONS: Biliary Tract Neoplasms
Keywords: biliary tract carcinoma; apatinib
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — apatinib

STUDY DESIGN:
Intervention Model Description: apatinib
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental): oral apatinib
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — oral apatinib 750mg qd

SUMMARY:
This is a phase II open-label, one-arm, single-center study of apatinib for eligible patients with advanced biliary tract carcinoma after the first-line treatment failure. A total of 55 patients is planned for enrollment. The time for enrollment is from Nov 2017 to Nov 2020, the the follow-up will be ended after Nov 2021. Patients in the study would receive oral apatinib 500-750mg qd until progression of disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age between 18 and 70 years
2. Histologically confirmed advanced biliary tract carcinoma (BTC) or metastatic BTC
3. Prior lack of response or intolerance to at least one chemotherapeutic regimens (including gemcitabine).
4. At least one measurable lesion as defined by RECIST 1.1
5. An Eastern Cooperative Oncology Group performance status of 0 to 2
6. Life expectancy ≥ 12 weeks
7. For those who received other anti-tumor treatment, the damage should have been restored, with the time interval from last dose of nitroso or mitomycin≥6 weeks and interval from last dose of other cytotoxic drugs, radiation or surgery (the wound should be healed completely) ≥4 weeks.
8. Acceptable hematologic, hepatic, and renal function within 7 days from screening： the blood ANC count≥1.5x109 /L; hemoglobin ≥ 9.0 g/dl，the blood platelet count≥80 x109 /L, total bilirubin < 1.5 x ULN, ALT and AST< 2.5 x ULN(< 5 x ULN for patients with live metastasis), serum creatinine≤1 x ULN，endogenous creatinine clearance rate >50ml/min
9. Women of reproductive age need to take effective contraceptive measures

Exclusion Criteria:

1. With other malignant tumor in 5 years，except for cured cervical carcinoma in situ or basal cell carcinoma.
2. Uncontrolled blood pressure on medication (140/90 mmHg); patients with > Grade 1 coronary heart disease, cardiac arrhythmias or cardiac dysfunction
3. Symptomatic brain or meningeal metastasis
4. History of uncontrolled seizures, central nervous system dysfunction or mental disorder
5. Uncontrolled pleural or peritoneal effusion
6. Undergoing dialysis
7. Severe or uncontrolled infection
8. With multiple factors that affecting oral administration
9. Abnormal coagulation function or those receiving thrombolytics or anticoagulants
10. Patients with tendency of gastrointestinal hemorrhage, including active peptic ulcer with fecal occult blood ++, hematemesis or melena within 3 months
11. Participation in other drug clinical trials within 4 weeks
12. Weight below 40kg
13. urine protein ≥2+

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
PFS | from the time signing of ICF until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  progression free survival

SECONDARY OUTCOMES:
OS | from the time signing of ICF until the date of death from any cause, assessed up to 48 months
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Weijian Guo, MD, Principal Investigator — Shanghai Cancer Hospital
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cereda S, Belli C, Rognone A, Mazza E, Reni M. Second-line therapy in advanced biliary tract cancer: what should be the standard? Crit Rev Oncol Hematol. 2013 Nov;88(2):368-74. doi: 10.1016/j.critrevonc.2013.05.010. Epub 2013 Jun 17. PMID 23786845
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Li J, Qin S, Xu J, Guo W, Xiong J, Bai Y, Sun G, Yang Y, Wang L, Xu N, Cheng Y, Wang Z, Zheng L, Tao M, Zhu X, Ji D, Liu X, Yu H. Apatinib for chemotherapy-refractory advanced metastatic gastric cancer: results from a randomized, placebo-controlled, parallel-arm, phase II trial. J Clin Oncol. 2013 Sep 10;31(26):3219-25. doi: 10.1200/JCO.2013.48.8585. Epub 2013 Aug 5. PMID 23918952
- [Background] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- [Background] Peng H, Zhang Q, Li J, Zhang N, Hua Y, Xu L, Deng Y, Lai J, Peng Z, Peng B, Chen M, Peng S, Kuang M. Apatinib inhibits VEGF signaling and promotes apoptosis in intrahepatic cholangiocarcinoma. Oncotarget. 2016 Mar 29;7(13):17220-9. doi: 10.18632/oncotarget.7948. PMID 26967384
- [Derived] Wang C, Huang M, Geng Q, Li W, Chang J, Tang W, Guo W. Apatinib for patients with metastatic biliary tract carcinoma refractory to standard chemotherapy: results from an investigator-initiated, open-label, single-arm, exploratory phase II study. Ther Adv Med Oncol. 2021 Aug 31;13:17588359211039047. doi: 10.1177/17588359211039047. eCollection 2021. PMID 34484431